CLINICAL TRIAL: NCT05158166
Title: DaxibotulinumtoxinA Injection for Treatment of Adductor Spasmodic Dysphonia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-33778
Record Dates: First submitted 2021-11-19; First posted 2021-12-15 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Adductor Spasmodic Dysphonia; Voice Disorders; Spasmodic Dysphonia
Keywords: adductor spasmodic dysphonia
MeSH Terms: conditions — Voice Disorders; Dysphonia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of Daxi (Experimental): Injectible daxibotulinumtoxinA (DAXI, Revance Therapeutics Inc., Newark, CA) is an investigational botulinum toxin type A which has been shown in large clinical trials to provide safe, effective treatment for glabellar lines and cervical dystonia and may offer longer-lasting results when compared with onabotulinumtoxinA. Dosage will be same number of units as prior Botox A dose.
  Interventions: Drug: DaxibotulinumtoxinA

INTERVENTIONS:
Drug: DaxibotulinumtoxinA — This is a long-acting alternative to traditional Botox A treatment.
  Other Names: DAXI

SUMMARY:
Spasmodic Dysphonia (SD) is a neurologic condition causing inappropriate contraction of the laryngeal musculature, leading to abnormal voicing. The three types (adductor, abductor, and mixed) affect varying muscle groups which produce characteristic voice patterns. The vast majority of patients with SD have adductor type, which impacts the lateral cricoarytenoid and thyroarytenoid muscle complex. While many treatment modalities have been investigated, the most effective treatment is botulinum toxin injection to these muscle groups, performed transcervically with or without electromyography (EMG) guidance. Patients undergoing this treatment typically require re-injection every 3 months. Due to its specialized nature, the laryngeal injections are not performed routinely outside of academic medical centers; thus, patients may come from a distance to receive this treatment. Both due to the significant impact on voice quality when the injections wear off and the sometimes challenging access to treatment, a longer-acting agent is desired.

Injectible daxibotuliumtoxinA (DAXI, Revance Therapeutics Inc., Newark, CA) has been shown in large clinical trials to provide safe, effective treatment for glabellar lines and cervical dystonia and may offer a longer-lasting result when compared with onabotulinumtoxinA.

Thus, a study examining the effect of DAXI for patients with adductor spasmodic dysphonia is proposed. This study aims to assess the efficacy of DAXI for transcervical laryngeal injection in patients with adductor spasmodic dysphonia.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18
* diagnosis of adductor spasmodic dysphonia
* previous successful treatment with BotoxA
* stabilized dose for last 3 treatments

Exclusion Criteria:

* age less than 18
* exclusively having other neurologic conditions such as:

  * abductor spasmodic dysphonia
  * ALS
  * Multiple sclerosis
  * Parkinson's disease
  * Essential tremor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
Our primary outcome is the difference in VHI-10 score at 6 weeks after injection with DAXI. | 6 weeks
  This will be determined using a paired t-test with subjects pre-treatment VHI-10 scores as a control.

SECONDARY OUTCOMES:
A secondary outcome will be comparing the duration of effect of DAXI with patients' prior Botox treatment. | Up to 1 year
  Specifically, we will determine the median time to baseline VHI-10 after treatment with DAXI and produce a Kaplan-Meier curve to illustrate the duration of clinical benefit.

CONTACTS AND LOCATIONS:
Overall Officials: Clark Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carruthers J, Solish N, Humphrey S, Rosen N, Muhn C, Bertucci V, Swift A, Metelitsa A, Rubio RG, Waugh J, Quiring J, Shears G, Carruthers A. Injectable DaxibotulinumtoxinA for the Treatment of Glabellar Lines: A Phase 2, Randomized, Dose-Ranging, Double-Blind, Multicenter Comparison With OnabotulinumtoxinA and Placebo. Dermatol Surg. 2017 Nov;43(11):1321-1331. doi: 10.1097/DSS.0000000000001206. PMID 28614091
- [Background] Jankovic J, Truong D, Patel AT, Brashear A, Evatt M, Rubio RG, Oh CK, Snyder D, Shears G, Comella C. Injectable DaxibotulinumtoxinA in Cervical Dystonia: A Phase 2 Dose-Escalation Multicenter Study. Mov Disord Clin Pract. 2018 Apr 26;5(3):273-282. doi: 10.1002/mdc3.12613. eCollection 2018 May-Jun. PMID 30009213
- [Background] Carruthers JD, Fagien S, Joseph JH, Humphrey SD, Biesman BS, Gallagher CJ, Liu Y, Rubio RG; SAKURA 1 and SAKURA 2 Investigator Group; SAKURA 1 and SAKURA 2 Investigator Group includes the following. DaxibotulinumtoxinA for Injection for the Treatment of Glabellar Lines: Results from Each of Two Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Studies (SAKURA 1 and SAKURA 2). Plast Reconstr Surg. 2020 Jan;145(1):45-58. doi: 10.1097/PRS.0000000000006327. PMID 31609882
- [Background] Stone HF, Zhu Z, Thach TQ, Ruegg CL. Characterization of diffusion and duration of action of a new botulinum toxin type A formulation. Toxicon. 2011 Aug;58(2):159-67. doi: 10.1016/j.toxicon.2011.05.012. Epub 2011 May 31. PMID 21658400
- [Background] Rumbach A, Aiken P, Novakovic D. RETRACTED: Outcome Measurement in the Treatment of Spasmodic Dysphonia: A Systematic Review of the Literature. J Voice. 2019 Sep;33(5):810.e13-810.e39. doi: 10.1016/j.jvoice.2018.03.011. Epub 2018 Apr 11. PMID 29655932 (Retraction: PMID 33678307 J Voice. 2021 Mar;35(2):331)